CLINICAL TRIAL: NCT06456931
Title: Comparing the Efficacy of Traditional Buddhist Mindfulness Training Versus Secular Mindfulness-based Cognitive Therapy for Residual Depressive Symptoms in Patients With Depressive Disorders: a Pilot Randomized Controlled Trial
Brief Title: A Pilot Study Comparing the Efficacy of Traditional Buddhist Mindfulness Training Versus Secular Mindfulness-based Cognitive Therapy for Patients Having Residual Depressive Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anuradha Baminiwatta (Other)
Collaborators: Curtin University (Other); University of Melbourne (Other)
Responsible Party: Sponsor-Investigator, Anuradha Baminiwatta, Lecturer, University of Kelaniya
Organization: University of Kelaniya (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P/18/02/2024
Record Dates: First submitted 2024-05-29; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Depression Moderate; Depression Mild
Keywords: mindfulness; depression; religiosity
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: As the study involves two psychological/behavioural interventions, it will not be possible to mask the participants, care providers or the investigators. However, most outcomes are based on self-report ratings, and the outcome at the end of the intervention (relapse of depression) will be assessed using telephone interviews by investigators blind to the participant's study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Buddhist mindfulness training (Experimental): This involves an 8-week program with weekly 2-hour sessions, and daily home practice of comparable duration to MBCT, conducted in groups of 15 participants. Sessions will be conducted by a lay mindfulness trainer inside a conference hall. Meditation practice will include sitting meditation, walking meditation, and loving-kindness meditation. In addition to meditation practice, sessions will involve teaching and discussing concepts related to mindfulness from the Pali Canon, placed within the context of fundamental principles of Buddhism. Anecdotes from Buddhist literature will also be used. Additionally, the participants will be given the opportunity to engage in religious rituals of their preference during the sessions. Participants will be encouraged to engage in meditation, along with preferred religious activities for at least 40 minutes a day.
  Interventions: Behavioral: Traditional Buddhist mindfulness
- Secular mindfulness based cognitive therapy (Active Comparator): Secular MBCT groups (each consisting of 15 participants) will undergo the manualized 8-week MBCT program (Segal et al., 2002). Weekly 2-hour sessions will be conducted inside a conference hall at the Faculty of Medicine, University of Kelaniya by the principal investigator who is a senior registrar in psychiatry with over 6 years of personal experience in mindfulness practice. Daily home practice of 40 minutes will be recommended. Guided meditation recordings made in Sinhalese will be provided for home practice. Some cognitive behavioural exercises will be prescribed as part of homework (e.g., Pleasant and Unpleasant Events Calendars).
  Interventions: Behavioral: secular mindfulness based cognitive therapy

INTERVENTIONS:
Behavioral: Traditional Buddhist mindfulness — Details are provided in the arm/group descriptions.
  Arms: Traditional Buddhist mindfulness training
Behavioral: secular mindfulness based cognitive therapy — Details are provided in the arm/group descriptions.
  Arms: Secular mindfulness based cognitive therapy

SUMMARY:
This interventional study is conducted with the goal of comparing the efficacy of traditional Buddhist mindfulness training versus secular mindfulness based cognitive therapy among patients with depressive disorders. We are also interested in studying how these interventions compare in terms of preventing further relapses of depression. Additionally, this study aims to identify factors that influence the efficacy of this intervention, such as self-report mindfulness, self-compassion, and religiosity.

DETAILED DESCRIPTION:
This study has the following objectives:

1. To investigate whether traditional Buddhist mindfulness training is non-inferior to secular MBCT in reducing depressive symptoms and improving psychological wellbeing (primary outcomes)
2. To compare the effectiveness of the two interventions on self-compassion, mindfulness, and spirituality/religiosity (secondary outcomes)
3. To investigate whether self-compassion, mindfulness, and spirituality/religiosity mediate the effectiveness of the interventions
4. To investigate whether baseline spirituality/religiosity moderates the effectiveness of the interventions
5. To compare the effectiveness of the two interventions in preventing depressive relapse over 6 months and 12 months.

This will be a parallel group, randomized controlled trial conducted at Colombo North Teaching Hospital (CNTH), and the Faculty of Medicine, University of Kelaniya and involves interventions conducted over 4 months, followed by 12 months of follow-up. Patients with a history of depressive disorder will be recruited from the Psychiatry Clinic, Colombo North Teaching Hospital. Sample size, calculated for a non-inferiority trial design, is 30 in each group. Simple randomization and allocation concealment using sequentially numbered, opaque, sealed envelopes will be used. Both groups will undergo interventions over 8 weeks, with weekly 2-hour sessions. One group will undergo the novel intervention, i.e., traditional Buddhist mindfulness training. The other group will undergo MBCT. Primary outcomes will be depressive symptom severity (Beck Depression Inventory-II), Psychological wellbeing (WHO-5 Wellbeing Index), and the depressive relapse rate at 6 months and 1 year after completion of intervention. Secondary outcomes include mindfulness (Six-Facet Mindfulness Questionnaire), Self-compassion (Self-compassion scale - short form), Spirituality/religiosity (BENEFIT scale), and Acceptability/feasibility. To establish non-inferiority, the 95% CI of the mean difference will be compared against the non-inferiority margin. Moderator and mediation analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Buddhist faith (Only Buddhists are selected as one of the interventions involves Buddhist teachings, and any recruited participant has a probability of being enrolled in the Buddhist mindfulness intervention)
* A history of one or more episodes of moderate or severe depression
* Currently having BDI-II score > 13, i.e., mild to moderate depressive symptoms

Exclusion Criteria:

* Currently having a severe depressive episode, according to the Composite International Diagnostic Interview (CIDI) Sinhalese version
* Currently having moderate to severe suicidal ideation (according to CIDI)
* Recent changes in antidepressant medication
* Unable to understand and communicate in Sinhalese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptom severity | Baseline (T0), Post-intervention (T1) 8 weeks from baseline
  Beck Depression Inventory -II Score
Psychological wellbeing | Baseline (T0), Post-intervention (T1) 8 weeks from baseline
  WHO Wellbeing Index - 5 score
Relapses of depression | At 6 months and 1 year after completion of intervention
  Depressive relapse rate assessed using Composite International Diagnostic Interview

SECONDARY OUTCOMES:
Self-report mindfulness | Baseline (T0), Post-intervention (T1) 8 weeks from baseline
  20-item Six-Facet Mindfulness Questionnaire - Sinhala (Baminiwatta et al. 2022)
Self-compassion | Baseline (T0), Post-intervention (T1) 8 weeks from baseline
  12-item Self-compassion scale - short form - Sinhala ( De Zoysa et al., 2021)
Spirituality/religiosity | Baseline (T0), Post-intervention (T1) 8 weeks from baseline
  6-item BENEFIT scale - Sinhala (Xue et al., 2016)

OTHER OUTCOMES:
Acceptability of the intervention | Post-intervention (T1) 8 weeks from baseline
  measured using two items: Item 1 will ask participants to rate their overall satisfaction with the intervention using a 10-point Likert scale ranging from 1 (quite dissatisfied) to 10 (very satisfied). Item 2 will ask participants to rate how helpful they believed the intervention was for them on a scale from 1 (not at all helpful) to 10 (very helpful).
Feasibility of the intervention | Post-intervention (T1) 8 weeks from baseline
  Session attendance (i.e., the total number of weekly sessions attended); home practice completion (i.e., number of days that home practice was completed); and retention rates will be used as indicators of feasibility. Home practice will be assessed using a homework record form over the 8-week intervention period. Retention rate will be operationalized as the percentage of enrolled participants who complete the primary outcome assessment, and attend at least 4 out of the 8 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Baminiwatta, MBBS, MD, Principal Investigator — University of Kelaniya
Locations (1):
- Colombo North Teaching Hospital, Ragama, Gampaha, Sri Lanka

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared publicly on Figshare.
Time Frame: Prior to the submission of the study findings to a journal
Access Criteria: Public